CLINICAL TRIAL: NCT06252376
Title: Effects of Blood Pressure on Cognition and Cerebral Hemodynamics in Parkinson's Disease
Brief Title: Effects of Blood Pressure on Cognition and Cerebral Hemodynamics in PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Katie Longardner, Assistant Clinical Professor of Health Sciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 210738a
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease; Orthostatic Hypertension; Cognitive Change; Cognitive Impairment; Cognitive Decline
Keywords: Parkinson's disease; Blood pressure; Blood flow; Cognition; fNIRS
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine cognitive testing first (Experimental): Participants will undergo a computerized cognitive battery in the supine position, followed by a similar battery with alternate test versions in the upright position while on a head-up tilt table.
  Interventions: Diagnostic Test: Head-up tilt table
- Upright cognitive testing first (Experimental): Participants will undergo a computerized cognitive battery in the upright position, followed by a similar battery with alternate test versions in the supine position while on a head-up tilt table.
  Interventions: Diagnostic Test: Head-up tilt table

INTERVENTIONS:
Diagnostic Test: Head-up tilt table — Different versions of cognitive assessments will be administered in the supine and upright positions while the participant is on the tilt table.

SUMMARY:
The goal of clinical trial is to learn about how blood pressure fluctuations affect cognitive performance (thinking abilities) and brain blood flow in persons with Parkinson's disease with and without orthostatic hypotension (low blood pressure when standing). The main questions it aims to answer are:

* Is there a certain level of blood pressure that correlates with change in cognitive performance while upright?
* Is there a certain level of change in brain blood flow that correlates with change in cognitive performance when upright?
* How does cognitive performance differ between persons with Parkinson's disease that have orthostatic hypotension and those without orthostatic hypotension?
* How does cognitive performance differ between the supine (laying down) and upright positions?
* How do blood pressure and brain blood predict changes in cognitive performance over two years?

Participants in this study will undergo the following procedures:

* Complete a screening visit with questionnaires, medical history, physical exam, and head-up tilt-table test.
* Attend one baseline study visit, during which they will undergo a battery of computerized cognitive tests repeated twice: once while laying down and once while upright on a tilt table. Simultaneously, during the experiments we will measure blood pressure using a wrist-worn device and inflatable arm cuff and will measure brain blood flow using functional near-infrared spectroscopy (fNIRS), a non-invasive device that uses light sensors to detect changes in brain blood flow.
* Attend one two-year follow-up visit, during which they will repeat a battery of computerized cognitive tests repeated twice: once while laying down and once while upright on a tilt table. During this visit, like before, we will measure blood pressure using a wrist-worn device and inflatable arm cuff and will measure brain blood flow using functional near-infrared spectroscopy (fNIRS).

Researchers will compare participants with Parkinson's disease with and without orthostatic hypotension in the laying down and upright positions to see if there are changes in thinking abilities between these groups.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease worldwide and causes disabling non-motor symptoms that include cognitive impairment and low blood pressure (BP) on standing, called orthostatic hypotension (OH). About 30-50% of people with PD have OH; cognitive impairment is also common in PD and has several causes. OH is associated with cognitive impairment in PD, but it is unknown to what extent OH could be a treatable risk factor for cognitive decline. People with PD and OH can experience sudden temporary cognitive dysfunction when upright, suggesting that OH-related drops in BP can transiently reduce blood flow to the brain. In PD, OH also correlates strongly with long-term cognitive decline, predicting a 7-times higher risk of dementia. But it is unclear to what extent episodic cerebral hypoperfusion from OH - even if asymptomatic - contributes to ischemic brain damage that impacts long-term cognitive impairment in PD, which is a critical knowledge gap.

This project's objective is to determine how BP affects positional cognitive performance and brain blood flow in PD. We hypothesize that in person with PD patients with OH, but not those without OH, a critical threshold of cerebral hypoperfusion correlates with acute, temporary cognitive deficits when upright compared to supine and contributes to chronic cognitive decline.

The proposed experiments will close the existing knowledge gaps by determining the associations between BP and cerebral hemodynamics (brain blood flow) with cognitive performance. Experiments will be performed at baseline and repeated at two years. Sixty non-demented individuals with PD with OH (n=30) and without OH (n=30) will complete a computerized battery of cognitive tests in the supine and upright positions on a tilt table while undergoing simultaneous, non-invasive, continuous monitoring of BP and brain hemodynamics using functional near-infrared spectroscopy (fNIRS). Aim 1 will determine how BP relates to cognitive performance while supine and while upright. Aim 2 will use fNIRS to determine how cerebral hemodynamics (fNIRS) relate to cognitive performance and BP. Aim 3 will repeat the baseline assessments at a two-year follow-up visit to determine which BP and fNIRS measures are most associated with cognitive decline. We will compare these outcomes in participants with and without OH. This study will yield novel data about the short-term and long-term effects of low BP on cognitive performance and brain hemodynamics. Improving understanding of how BP affects cognition in PD will advance knowledge toward developing treatment targets to reverse, prevent, or delay OH-related cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease (PD) using the Movement Disorders Society (MDS) Clinical Diagnostic Criteria (Postuma, 2015)
* Age least 50 years old
* Hoehn & Yahr (H&Y) stages I to III (early to moderate stage PD)
* Proficiency in the English language (native English speaker level)

Exclusion Criteria:

* Any involuntary movements (i.e., tremor or dyskinesia) greater than 3 cm in amplitude, since the motion artifact can interfere with BP monitor cuff
* Taking antihypertensive medications or alpha-adrenergic blocking medications since these can cause hypotension.
* Dementia (including PD dementia (Emre, 2007) characterized by either Dementia Rating Scale 2 (DRS-2) score) 124 or less or clinical evidence of impaired instrumental activities of daily living
* History of deep brain stimulation (DBS) surgery
* Any unstable, active medical problem, e.g., decompensated heart failure, liver failure, etc.
* Moderate or severe carotid artery stenosis (according to North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria (Ferguson, 1999)
* History of cerebral infarction or hemorrhage
* Uncontrolled diabetes or any other systemic disease that causes autonomic failure
* Any terminal illness with life expectancy less than 2 years
* Illiteracy
* Impairment of hearing or vision that is not corrected by devices (e.g., hearing aids or glasses)
* Currently pregnant (will be confirmed with a urine pregnancy screening test in people of child-bearing potential)
* Any other condition, which, in the opinion of the investigator, could place the participant at increased risk (e.g., substance abuse)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Verbal fluency score (number of words generated in one minute) | 24 months
  Participant names as many words from a prompt as possible in one minute. Minimum: 0; Maximum: N/A; higher is better
Blood pressure (mmHg) | 24 months
  Participants' blood pressure will be measured during the visit.
Oxygenated hemoblobin change from baseline | 24 months
  Functional near-infrared spectroscopy will measure relative changes in oxygenated hemoglobin during cognitive testing.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Longardner K, Bayram E, Litvan I. Orthostatic Hypotension Is Associated With Cognitive Decline in Parkinson Disease. Front Neurol. 2020 Sep 2;11:897. doi: 10.3389/fneur.2020.00897. eCollection 2020. PMID 32982926
- [Background] Freeman R, Illigens BMW, Lapusca R, Campagnolo M, Abuzinadah AR, Bonyhay I, Sinn DI, Miglis M, White J, Gibbons CH. Symptom Recognition Is Impaired in Patients With Orthostatic Hypotension. Hypertension. 2020 May;75(5):1325-1332. doi: 10.1161/HYPERTENSIONAHA.119.13619. Epub 2020 Mar 30. PMID 32223377
- [Background] Gibbons CH, Schmidt P, Biaggioni I, Frazier-Mills C, Freeman R, Isaacson S, Karabin B, Kuritzky L, Lew M, Low P, Mehdirad A, Raj SR, Vernino S, Kaufmann H. The recommendations of a consensus panel for the screening, diagnosis, and treatment of neurogenic orthostatic hypotension and associated supine hypertension. J Neurol. 2017 Aug;264(8):1567-1582. doi: 10.1007/s00415-016-8375-x. Epub 2017 Jan 3. PMID 28050656
- [Background] Udow SJ, Robertson AD, MacIntosh BJ, Espay AJ, Rowe JB, Lang AE, Masellis M. 'Under pressure': is there a link between orthostatic hypotension and cognitive impairment in alpha-synucleinopathies? J Neurol Neurosurg Psychiatry. 2016 Dec;87(12):1311-1321. doi: 10.1136/jnnp-2016-314123. Epub 2016 Sep 9. PMID 27613160
- [Background] McDonald C, Newton JL, Burn DJ. Orthostatic hypotension and cognitive impairment in Parkinson's disease: Causation or association? Mov Disord. 2016 Jul;31(7):937-46. doi: 10.1002/mds.26632. Epub 2016 Apr 19. PMID 27091624
- [Background] Poda R, Guaraldi P, Solieri L, Calandra-Buonaura G, Marano G, Gallassi R, Cortelli P. Standing worsens cognitive functions in patients with neurogenic orthostatic hypotension. Neurol Sci. 2012 Apr;33(2):469-73. doi: 10.1007/s10072-011-0746-6. Epub 2011 Sep 6. PMID 21894556
- [Background] Centi J, Freeman R, Gibbons CH, Neargarder S, Canova AO, Cronin-Golomb A. Effects of orthostatic hypotension on cognition in Parkinson disease. Neurology. 2017 Jan 3;88(1):17-24. doi: 10.1212/WNL.0000000000003452. Epub 2016 Nov 30. PMID 27903817
- [Background] Pinti P, Tachtsidis I, Hamilton A, Hirsch J, Aichelburg C, Gilbert S, Burgess PW. The present and future use of functional near-infrared spectroscopy (fNIRS) for cognitive neuroscience. Ann N Y Acad Sci. 2020 Mar;1464(1):5-29. doi: 10.1111/nyas.13948. Epub 2018 Aug 7. PMID 30085354
- [Background] Palma JA, Gomez-Esteban JC, Norcliffe-Kaufmann L, Martinez J, Tijero B, Berganzo K, Kaufmann H. Orthostatic hypotension in Parkinson disease: how much you fall or how low you go? Mov Disord. 2015 Apr 15;30(5):639-45. doi: 10.1002/mds.26079. Epub 2015 Feb 12. PMID 25678194
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Kaufmann H, Malamut R, Norcliffe-Kaufmann L, Rosa K, Freeman R. The Orthostatic Hypotension Questionnaire (OHQ): validation of a novel symptom assessment scale. Clin Auton Res. 2012 Apr;22(2):79-90. doi: 10.1007/s10286-011-0146-2. Epub 2011 Nov 2. PMID 22045363
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984